CLINICAL TRIAL: NCT07256782
Title: A Phase Ib/II, Open-label, Multi-center Study to Evaluate Safety, Tolerability, Pharmacokinetics and Efficacy of Intravenous Administration of QLC5508 in Combination With Other Anti-tumor Agents in Patients With Advanced Solid Tumors
Brief Title: A Study of QLC5508 Combinations in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLC5508-201
Record Dates: First submitted 2025-09-28; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Cisplatin; Carboplatin; Paclitaxel; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- QLC5508 and QL1706 (Experimental)
  Interventions: Drug: QLC5508; Drug: QL1706
- QLC5508, QL1706 and Cisplatin/ Carboplatin (Experimental)
  Interventions: Drug: QLC5508; Drug: QL1706; Drug: Cisplatin/ Carboplatin
- QLC5508 and QL2107 (Experimental)
  Interventions: Drug: QLC5508; Drug: QL2107
- QLC5508, QL2107 and 5-fluorouracil (5-FU) (Experimental)
  Interventions: Drug: QLC5508; Drug: QL2107; Drug: 5-fluorouracil (5-FU)
- QLC5508, QL2107 and Paclitaxel (Experimental)
  Interventions: Drug: QLC5508; Drug: QL2107; Drug: Paclitaxel
- QLC5508, Oxaliplatin, 5-fluorouracil (5-FU) and leucovorin (Experimental)
  Interventions: Drug: QLC5508; Drug: 5-fluorouracil (5-FU); Drug: Oxaliplatin

INTERVENTIONS:
Drug: QLC5508 — 2.4 mg/kg and 2.0 mg/kg, Q3W/Q2W,administered as an IV infusion
  Other Names: MHB088C
Drug: QL1706 — 5 mg/kg ,Q3W,administered as an IV infusion
  Other Names: Iparomlimab and Tuvonralimab，PSB205
  Arms: QLC5508 and QL1706; QLC5508, QL1706 and Cisplatin/ Carboplatin
Drug: Cisplatin/ Carboplatin — Cisplatin(75 mg/m2; Q3W) / Carboplatin（AUC 5 mg/mL/min; Q3W）,administered as an IV infusion
  Arms: QLC5508, QL1706 and Cisplatin/ Carboplatin
Drug: QL2107 — 200 mg, Q3W,administered as an IV infusion
  Arms: QLC5508 and QL2107; QLC5508, QL2107 and 5-fluorouracil (5-FU); QLC5508, QL2107 and Paclitaxel
Drug: Paclitaxel — 175 mg/m2, Q3W,administered as an IV infusion
  Arms: QLC5508, QL2107 and Paclitaxel
Drug: 5-fluorouracil (5-FU) — 800 mg/m2,Q3W(arm:QLC5508, QL2107 and 5-FU),administered as an IV infusion;1200 mg/m2, Q2W(arm:QLC5508, Oxaliplatin, 5-FU,and leucovorin),administered as an IV infusion
  Arms: QLC5508, Oxaliplatin, 5-fluorouracil (5-FU) and leucovorin; QLC5508, QL2107 and 5-fluorouracil (5-FU)
Drug: Oxaliplatin — 30 mg/m2, Q2W,administered as an IV infusion
  Arms: QLC5508, Oxaliplatin, 5-fluorouracil (5-FU) and leucovorin

SUMMARY:
QLC5508 is a fully humanized IgG1 antibody-drug conjugate (ADC) which specifically binds to B7-H3, a target wildly expressed on solid tumor cells. The objectives of this study are to investigate the safety, tolerability, pharmacokinetics and anti-tumor activity of QLC5508 in combination with other anti-cancer agents in patients with advanced solid tumor patients.

DETAILED DESCRIPTION:
This is a phase Ib/II, open-label, multi-center, dose-escalation and expansion in Chinese subjects with advanced solid tumors. This study is in design allowing assessment of safety, tolerability, pharmacokinetics and anti-tumor activity of QLC5508 in combination with other anti-cancer agents.

The target population of dose escalation part is patients have progressed on or intolerant to available standard therapies, and the dose expansion part will enroll patients who have not received prior treatment for advanced/metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at screening;
* Histologically or cytologically confirmed advanced solid tumors:

Dose escalation part will enroll participants who have progressed on or are intolerant to available standard therapies.

Dose expansion part will enroll participants who have not received prior treatment for advanced/metastatic diseases.

* At least one measurable target lesion according to RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0~1
* Life expectancy ≥12 weeks
* Female or male participants should be willing to use appropriate contraceptive measures throughout the study;
* Female participants should have a negative blood pregnancy test within 7 days prior to the first dose or have evidence of non-childbearing potential;
* A signed written Informed Consent Form

Exclusion Criteria:

* . Received or undergoing any of the following treatment:

  1. Previous or current treatment with B7-H3 targeted therapy
  2. Previous or current treatment with topoisomerase I inhibitors
  3. Previous treatment with cytotoxic chemotherapy, investigational agents, traditional Chinese medicine with an anti-tumor indication and antitumor drugs within 14 days prior to the first dose
  4. Previous treatment with macromolecular antitumor drugs within 28 days prior to the first dose

  f. Radiotherapy with a limited field of radiation within 2 weeks prior to the first dose; or more than 30% of the bone marrow irradiation, or large-scale radiotherapy within 4 weeks prior to the first dose e. Pleural effusion or ascites requiring clinical intervention; or presence of pericardial effusion f. Major surgery within 4 weeks prior to the first dose g. Brain metastases; leptomeningeal or brainstem metastases; or spinal cord compression
* Unresolved AEs ≥ Grade 2 (CTCAE v5.0) from prior therapy except for alopecia and residual neuropathy
* Previous or concurrent primary malignancies
* Inadequate bone marrow reserve or organ dysfunction
* Evidence of cardiovascular risk
* Evidence of current severe or uncontrolled systemic diseases
* Severe infection within 4 weeks prior to the first dose; or uncontrolled active infection at screening
* Known or suspected interstitial lung disease; or other moderate to severe pulmonary diseases that significantly impair respiratory function and may interfere with the detection or management of drug-related pulmonary toxicity
* High risk of gastrointestinal or abdominal bleeding 10. Gastrointestinal diseases of clinical significance within 3 months prior to the first dose
* History of severe neuropathy or mental disorders
* History of severe hypersensitivity reaction, severe infusion reaction or idiosyncrasy to drugs chemically related to QLC5508 or any of the components of QLC5508
* Unlikely to comply with study procedures and requirements in the opinion of the investigator
* Any disease or condition that, in the opinion of the investigator, would compromise participant safety or interfere with study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) for combination-treatments (Phase Ib) | Up to day 21 (Q3W combination) or day 28 (Q2W combination) from the first dose
  To determine the MTD for further evaluation of QLC5508 with other anti-cancer agents in participants with advanced solid tumors
Recommended Phase II Dose (RP2D) for combination-treatments (Phase Ib) | Up to day 21 (Q3W combination) or day 28 (Q2W combination) from the first dose
  To determine the RP2D for further evaluation of QLC5508 with other anti-tumor agents in participants with advanced solid tumors
Objective response rate (ORR) determined by investigators (Phase II) | Approximately 12 months
  ORR is defined as proportion of participants with best overall response of complete response (CR) and partial response (PR) [Confirmed CR/PR assessment require at least one repeat (4-6 weeks)] evaluated by investigator according to RECIST v1.1

SECONDARY OUTCOMES:
ORR determined by investigators (Phase Ib) | Approximately 12 months
  ORR is defined as proportion of participants with best overall response of CR and PR [Confirmed CR/PR assessment require at least one repeat (4-6 weeks)] evaluated by investigator according to RECIST v1.1
Disease control rate (DCR) determined by investigators (Phase Ib and II) | Approximately 12 months
  DCR is defined as proportion of participants with best overall response of CR, PR and stable disease (SD) evaluated by investigator according to RECIST v1.1 [Confirmed CR/PR assessment require at least one repeat (4-6 weeks)]
Duration of response (DOR) determined by investigators (Phase Ib and II) | Approximately 12 months
  DOR is defined as the period from the first occurrence of CR or PR to PD or death from any cause [Confirmed CR/PR assessment require at least one repeat (4-6 weeks)]
Progression-free survival (PFS) determined by investigators (Phase Ib and II) | Approximately 12 months
  PFS is defined as the time from the first dose to PD or death from any cause.
Overall survival (OS) (Phase Ib and II) | Approximately 24 months
  OS is defined as the time from the first dose to death from any cause
Incidence and severity of adverse events (AEs) (Phase II) | From the first dose through 90 days post end of treatment
  Any untoward medical occurrence in a clinical study participant, which may manifest as symptoms, signs, diseases, or laboratory abnormalities, are assessed by investigator according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), v5.0
Observed maximum plasma concentration (Cmax) of QLC5508 in advanced solid tumor (Phase Ib and II) | From pre-dose to study completion, approximately 24 months
  Cmax will be obtained after administration of the first dose of QLC5508
Time to reach maximum plasma concentration (Tmax) of QLC5508 (Phase Ib) | From pre-dose to study completion, approximately 24 months
  Tmax will be obtained after administration of the first dose of QLC5508
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) following the first dose of QLC5508 (Phase Ib) | From pre-dose to study completion, approximately 24 months]
  Area under the plasma concentration versus time curve from time zero to the last sampling time when the concentration was no less than the lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Observed maximum plasma concentration (Cmax) of QL1706 in advanced solid tumor (Phase Ib and II) | From pre-dose to study completion, approximately 24 months
  Cmax will be obtained after administration of the first dose of QL1706
Observed maximum plasma concentration (Cmax) of QL2107 in advanced solid tumor (Phase Ib and II) | From pre-dose to study completion, approximately 24 months
  Cmax will be obtained after administration of the first dose of QL2107
Percentage of participants with antibodies to QLC5508 in serum (Phase Ib and II) | From pre-dose to study completion, approximately 24 months
  Serum samples were collected for the determination of anti-drug antibody (ADA) at designated time points.
Percentage of participants with antibodies to QL1706 in serum (Phase Ib and II) | From pre-dose to study completion, approximately 24 months
  Serum samples were collected for the determination of ADA at designated time points

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China